CLINICAL TRIAL: NCT07078097
Title: "A Heritage of Healing: Traditional Song and Its Anxiety-Mitigating Effects During Pregnancy"
Brief Title: Healing Sounds for Pregnant Women: Sape' Dayak Music and Anxiety Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Polytechnic of Palangka Raya (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 470/II/KE.PE/2025; HK.02.03/XLI/1802/2025 (Other: Health Polytechnic of Palangkaraya)
Record Dates: First submitted 2025-06-22; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Anxiety
Keywords: pregnancy; anxiety; music therapy; lullabies; traditional music; mental health
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study used a quasi-experimental design with a control group, meaning participants were not randomly assigned. Instead, assignment was based on the midwifery clinic attended: clinic A for the Sape' Dayak intervention group (IG) and clinic B for the Brahms' Lullaby control group (CG). A pre-test and post-test design was used, with anxiety levels measured by the Perinatal Anxiety Screening Scale (PASS) before and after the intervention. The intervention involved 20 minutes of music listening daily for three consecutive days. This was conducted in participants' homes for comfort and privacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG): Traditional Sape' Dayak Music (Experimental): Participants will listen to one Sape' Dayak song for 20 minutes daily over three consecutive days. This traditional Dayaknese song features pentatonic melodies known for creating a serene and emotionally relaxing environment, ideal for healing and anxiety relief. While listening through earphones, participants will be instructed to gently massage their abdomens and imagine their infants. The Sape' Dayak music has a slow rhythm, fluctuating between 80 to 85 beats per minute, which aligns with the normal heart rate. Sessions will be held in participants' homes for privacy, between 08:00 and 11:00 post-breakfast, ensuring no medical care or other distractions.
  To ensure participants compliance, the trackify music tracking app will be used, and research assistants will collect the time of playing from the app upon completion of the session.
  Interventions: Other: Traditional Sape' Dayak Music Listening
- Control Group (CG): Brahms' Lullaby Music Therapy (Active Comparator): Participants will listen to one preselected Johannes Brahms' Lullaby song for 20 minutes daily for three consecutive days. The lyrics typically express maternal love and tenderness for the fetus. Similar to the IG, participants will be instructed to gently touch their tummy and reflect on their unborn children while wearing earphones. The intervention will take place in their homes during the same morning hours, minimizing external influences. This standardized approach aims to avoid bias from personal music preferences.
  To ensure participants compliance, the trackify music tracking app will be used, and research assistants will collect the time of playing from the app upon completion of the session.
  Interventions: Other: Brahms' Lullaby Music Therapy

INTERVENTIONS:
Other: Traditional Sape' Dayak Music Listening — This intervention is distinguished by its use of the Sape' Dayak, a specific traditional musical instrument from East Kalimantan, Indonesia, known for its gentle, contemplative, and culturally significant sounds. The music utilizes pentatonic melodies that foster a serene and emotionally relaxing environment. Its distinct rhythm (80-85 beats per minute) is also a key feature. The intervention also incorporates a gentle abdominal massage and imagining the infant.
  Arms: Intervention Group (IG): Traditional Sape' Dayak Music
Other: Brahms' Lullaby Music Therapy — This intervention is distinguished by its use of a globally popular and well-known lullaby composed by Johannes Brahms. The lyrics typically revolve around themes of love and affection, expressing mothers' love and tenderness for their fetuses. Unlike the Sape' Dayak, the specific lullaby will be preselected by the researcher to ensure a homogeneous intervention, with personal lullaby preferences ignored to avoid bias. Participants also engage in gentle abdominal touching and reflection on their unborn children.
  Arms: Control Group (CG): Brahms' Lullaby Music Therapy

SUMMARY:
This study investigates whether listening to traditional Dayak Sape' music could reduce anxiety in pregnant women as effectively as traditional lullabies. The researchers will recruit 32 pregnant women and divide them into two groups: one listened to Sape' Dayak music, and the other listened to Brahms' Lullaby. Anxiety levels will be measured before and after the music interventions using the Perinatal Anxiety Screening Scale (PASS).

DETAILED DESCRIPTION:
Pregnancy is a wonderful experience, but it can also be a source of anxiety for many women owing to hormonal changes, body changes, and the prospect of motherhood. This anxiety is not just uncomfortable; it can have a substantial influence on both the mother's and the baby's health. Recognizing this, experts are increasingly turning at non-medical approaches to aid, and music therapy is gaining popularity due to its low side effects.

Music has long been used for relaxation in various cultures, and it has been shown to have an effect on our physiology, including hormone release. This study will look specifically at the possibility of the Sape' Dayak, a traditional Indonesian instrument, as a therapeutic tool. The Sape' is noted for its relaxing properties and has a significant cultural value for the Dayak people. It is frequently utilized in healing rituals and community activities. While its cultural significance is evident, its specific benefit in relieving anxiety in pregnant women has not been extensively researched.

The primary purpose of this study is to address that research gap. The study is seeking to determine whether listening to Sape' Dayak music may reduce anxiety levels in pregnant mothers as effectively as traditional lullabies. The study intends to encourage holistic health practices while also contributing to the preservation of cultural heritage.

The study is designed as a quasi-experiment, with a control group. Researchers will recruit 32 pregnant women in the third trimester (28-40 weeks) from midwifery clinics. Participants require to be at least 18 years old, have poor sleep quality (a PSQI score of 5 or above). They will be eliminated if they are more than 40 weeks pregnant, have a mental disorder that affects their view of reality, or are carrying twins.

The 32 respondents will be split into two groups of sixteen each. One group, the intervention group (IG), will listen traditional Sape' Dayak music. The control group (CG) will listen to Brahms' Lullaby. Participants in both groups will be told to lightly massage their abdomens and visualize their infants while listening to music through earbuds for 20 minutes a day for three days straight. The music sessions will be held in the participants' homes to ensure privacy and comfort, with doors and windows closed.

Anxiety levels will be measured using the Perinatal Anxiety Screening Scale (PASS) both before (pre-test) and after the music intervention. The PASS is a solid and useful measure for identifying anxiety symptoms unique to perinatal women. The PASS scores assist characterize anxiety as little, mild-moderate, or severe. The acquired data will be examined using statistical software to assess anxiety levels across and within groups.

ELIGIBILITY:
Inclusion Criteria:

1). Third trimester of pregnancy (28-40 weeks); 2). At least 20 years old; 3). Having a score on the Pittsburgh Sleep Quality Index (PSQI) score > 5, which indicates poor sleep quality; 3). Primiparous.

Exclusion Criteria:

1. . Beyond the 40th week of pregnancy;
2. . Having mental illness that caused hallucinations or altered perception of reality;

5). Having a twin pregnancy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The eligibility criteria and exclusion criteria refer to "women" and "mother/maternal" terms. This study's eligibility is limited by biological sex (females who are pregnant).
Enrollment: 32 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
The Perinatal Anxiety Screening Scale (PASS) | The anxiety levels of the participants will be assessed before the music intervention (pre-test) and after the music intervention (post-test). The post-test assessment will be conducted 20 minutes after the 3-day music intervention.
  The primary outcome measure is the level of anxiety in pregnant women, assessed using the Perinatal Anxiety Screening Scale (PASS). This self-report instrument consists of 31 items, with participants rating subjective anxiety on a Likert scale from 0 (not at all) to 3 (very much). The PASS will be administered before and after the music intervention. It identifies anxiety symptoms specific to perinatal women and includes four subscales: acute anxiety and adjustment; general concern and specific fears; perfectionism, control, and trauma; and social anxiety. The total score is the sum of individual item scores. A cut-off score of 26 indicates clinically significant anxiety, with categories of minimal (0-20), mild-moderate (21-26), and severe (>26) anxiety. The PASS is validated and reliable in both English and Bahasa versions.
The level of anxiety in pregnant women, assessed using the Perinatal Anxiety Screening Scale (PASS) | The anxiety levels of the participants will be assessed before the music intervention (pre-test) and after the music intervention (post-test). The post-test assessment will be conducted 20 minutes after the 3-day music intervention.
  The primary outcome measure is the level of anxiety in pregnant women, assessed using the Perinatal Anxiety Screening Scale (PASS). This self-report instrument consists of 31 items, with participants rating subjective anxiety on a Likert scale from 0 (not at all) to 3 (very much). The PASS will be administered before and after the music intervention. It identifies anxiety symptoms specific to perinatal women and includes four subscales: acute anxiety and adjustment; general concern and specific fears; perfectionism, control, and trauma; and social anxiety. The total score is the sum of individual item scores. A cut-off score of 26 indicates clinically significant anxiety, with categories of minimal (0-20), mild-moderate (21-26), and severe (>26) anxiety. The PASS is validated and reliable in both English and Bahasa versions.

CONTACTS AND LOCATIONS:
Overall Officials: Erina Eka Hatini, Master, Principal Investigator — Health Polytechnic of Palangkaraya
Locations (1):
- Midwifery clinics, Palangkaraya, Central Kalimantan, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The study intended to share anonymized Individual Participant Data (IPD), which included raw and processed data for all main and secondary results, demographic details, and information on how well participants followed the intervention, with all personal identifiers taken out. In addition to the IPD, the final approved versions of the study protocol and the statistical analysis plan (SAP) were shared. Anonymized versions of the participant informed consent form (ICF), which were the data collection instruments, were also provided.
  Data was shared with qualified researchers involved in this study. The removal of identification meant that all direct identifiers, like names, addresses, phone numbers, and exact times of birth, enrolment, or assessment, were taken away for good. Each participant's data was given a unique, nameless code so that it could be tracked within the removed dataset without giving separate the participant's name.
Supporting Information: SAP, ICF
Time Frame: De-identified IPD will be generally made available to qualified researchers within six months following the primary publication of the study's main results, and data access requests can be submitted from that point forward.
Access Criteria: The main way that data will be shared is through a safe, limited-access data repository. We share data using an encrypted storage medium after getting permission.
URL: https://polkesraya.ac.id/ppid/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-07-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT07078097/Prot_ICF_000.pdf